CLINICAL TRIAL: NCT06818630
Title: Enhanced Photoaging Reversal Efficacy and Safety of 755nm Alexandrite Picosecond Laser with Diffractive Lens Array (DLA) in Conjunction with Integrated Skin Care for Skin Quality Improvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: L'Oréal Taiwan Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: IRB-24-044-A2_LOREAL(CE/DD/24)
Record Dates: First submitted 2025-02-07; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Skin Quality Improvement
Keywords: picosecond laser; CE/DD/242

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental side (Experimental): The experimental side receiving a combination treatment of SkinCeuticals skincare products, regular moisturizing product, and sunscreen on one half of the face, following 755nm alexandrite picosecond laser with DLA.
  Interventions: Other: SkinCeuticals combination skin care products; Other: Regular skin care procedure
- Control side (Experimental): The control side receiving the regular moisturizing product and sunscreen on the corresponding half of the face, following 755nm alexandrite picosecond laser with DLA.
  Interventions: Other: Regular skin care procedure

INTERVENTIONS:
Other: SkinCeuticals combination skin care products — 1. CE Ferulic Serum,
  2. Discoloration Defense (3% Tranexamic Acid),
  3. Triple Lipid Restore 2:4:2
  Arms: Experimental side
Other: Regular skin care procedure — 1. Regular moisturizing product (Phyto Corrective Gel),
  2. sunscreen (Advanced Brightening UV Defense SPF50 PA++++)

SUMMARY:
This study evaluates enhanced photoaging reversal efficacy and safety of 755nm alexandrite picosecond laser with diffractive lens array (DLA) in conjunction with integrated skin care for skin quality improvement. It is a single-center, evaluator-blinded, randomized spilt-face design. It is expected to recruit 35 patients whose face with simple pigmentation and photoaging in Dr. Lin's Dermatology Clinic.

Each subject will receive both treatment and control procedures according to the side = 1:1 ratio randomly assigned in two spilt-face usage. One spilt-face side is undergoing the treatment procedure with combination skin care products (CE/DD/242), and regular moisturizing product and sunscreen (Phyto Corrective Gel and Advanced Brightening UV Defense SPF50 PA++++). Another spilt-face side is undergoing the control procedure: regular moisturizing product and sunscreen (Phyto Corrective Gel and Advanced Brightening UV Defense SPF50 PA++++). This study includes a total of 3 cycles of treatment (weeks 0-4, 4-8, and 8-12). After each cycle, the effect and satisfaction of the treatment were evaluated once (weeks 4, 8, and 12). For redness/swelling outcome, the self-reported effect will be collected by phone call, or being evaluated by visit within 3 day after additional visits (0w+3d, 4w+3d, and 8w+3d).

Generalized linear mixed models will be used to assess whether the patterns of change in the mean response/proportion of each endpoint over time are the same in the treatment procedure and the control procedure. Among the primary endpoint family, either one with statistically significant will meet the study success criteria. The endpoints include (1) Wrinkles (2) Ultraviolet spots (3) Brown spots (4) Texture (5) Red blood vessels (6) Pores (7) Porphyrin (8) Hydration (9) Elasticity (10) Physician's general assessment (12) Subject satisfaction. All statistical analysis will be implement in SAS 9.4 and STATA 18.

DETAILED DESCRIPTION:
Patients undergoing picosecond laser treatment experience skin sensitivity, compromised barrier function, increased water loss, and oxidative stress post-treatment. Inadequate postoperative care prolongs recovery and raises the risk of pigmentation issues or recurrence. Common postoperative care includes antioxidants, moisturizing sunscreen, skin whitening, spot lightening, and barrier repair treatments. Common post-procedure skincare products include (1) CE Serum (an antioxidant serum containing vitamin C, vitamin E, and ferulic acid), (2) DD Serum (a serum containing tranexamic acid, kojic acid, and niacinamide [vitamin B3], which helps reduce pigmentation), and (3) Sebum membrane repair cream [242 cream] (a newly formulated cream designed to restore the skin barrier function caused by aging). However, standardized post-picosecond laser care protocols are lacking, necessitating more clinical data and experience summaries.

This study seeks to assess the effectiveness and satisfaction of combining SkinCeuticals skin-care products (CE/DD/242) with 755nm alexandrite picosecond laser with diffractive lens array (DLA) for facial pigmentation and photoaging. It will be a prospective, single-center, evaluator-blinded, randomized spilt-face design trial. Thirty-five subjects will be recruited and randomly assigned to receive either the combined skincare products (CE/DD/242), and regular moisturizing product and sunscreen (Phyto Corrective Gel and Advanced Brightening UV Defense SPF50 PA++++) (treatment group) or regular moisturizing product and sunscreen alone (control group) following 755nm alexandrite picosecond laser with DLA. The study consists of three treatment cycles over 12 weeks, with assessments conducted at the end of each cycle. Evaluation indicators will be compared at 4, 8, and 12 weeks post-treatment to determine efficacy and satisfaction. Additionally, the redness within 3 day will be collected through phone call or visit at trial site. The study aims to explore the maintenance medical benefits of combining 755nm alexandrite picosecond laser with DLA in conjugated with SkinCeuticals skincare products for facial pigmentation and photoaging.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 25-65 years of age on the date of informed consent
* Fitzpatrick skin type II-V with pigmentation and photoaging on both sides of the face
* The severity of pigmentation and photoaging on both sides of the face is the same.
* Willing to receive picosecond laser treatment.
* Willing to follow the research requirements and cooperate with the process for follow-up visits.
* Subjects able to understand the written informed consent and willing to subject as evidenced by signing the informed consent

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or planning to conceive within one year.
* Subjects with active facial melasma.
* Those with a history of skin pigmentation disorders, such as pigmentation induced by hormonal factors (pregnancy, oral contraceptives).
* Subjects with autoimmune diseases, endocrine disorders, or liver diseases that lead to changes in skin color.
* Subjects who have used skin whitening agents, steroids, or photosensitive drugs within the past three months.
* Subjects who have undergone laser treatment within the past three months.
* Those who have contraindications to picosecond laser or the CE/DD/242 products, or are allergic to the ingredients in the skincare combination products.
* Subjects with facial infections or inflammation.
* Those planning to use other medications affecting skin color during the study or in-tending to undergo other laser treatments or sunbathing.
* Subjects currently participating in other clinical trials.
* Subjects deemed unsuitable for participation in this study after evaluation by the researchers.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-07-29 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
The change of wrinkles, ultraviolet spots, brown spots, texture, pores, porphyrin, redness, blood vessels, hydration | Weeks 0, 4, 8, and 12
  The scores for wrinkles, ultraviolet spots, brown spots, texture, pores, porphyrin, redness, blood vessels, and hydration are measured using the VISIA skin analysis system (Canfield Scientific, USA).
Improvement in hydration and elasticity | Weeks 0, 4, 8, and 12
  The score of hydration and elasticity are measured by Focuskin.
Physician Assessments | Weeks 0, 4, 8, and 12
  The assessments by physicians based on digital photographs of the subjects' faces, scored from 0 to 4.
Participant satisfaction | Weeks 4, 8, and 12
  A questionnaire will be used to assess the overall satisfaction of the subjects regarding the skin care products. The satisfaction levels are classified as: Very Satisfied, Satisfied, Unsatisfied, and Very Unsatisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Bright Skin Clinic, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No